CLINICAL TRIAL: NCT04956315
Title: Accuracy and Stability of a New Automatic Knee Arthrometer in Diagnosing Anterior Cruciate Ligament Rupture
Brief Title: Accuracy and Stability of a New Automatic Knee Arthrometer in Diagnosing ACL Rupture
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beihang University (Other)
Responsible Party: Sponsor
Other Study IDs: M2020263
Record Dates: First submitted 2021-06-27; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Knee Ligament; Laxity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Examiner effect group: Two examiners performed the test on one healthy subject with both devices for ten consecutive days. We measured the AD of both knees and calculated the ADD of every test. We evaluated the contralateral-side effect by comparing the AD standard deviations of each knee with both devices, and compared the average ADD tested by different examiners with the same device, to estimate examiner effect.
  Interventions: Diagnostic Test: Side-to-side difference (reproducibility)
- Method effect group: The experienced examiner performed tests on 20 healthy subjects using both devices. The means and standard deviations of both knees were calculated. We examined the difference in measurements using each device to determine the method effect.
  Interventions: Diagnostic Test: Side-to-side difference (availability)
- Equipment effectiveness group: The experienced examiner performed tests on 200 ACL ruptureand 200 healthy subjects using each device. Effectiveness was analyzed using 1.5 mm and 3 mm threshold values in ACL tears.
  Interventions: Diagnostic Test: Side-to-side difference (Accuracy)

INTERVENTIONS:
Diagnostic Test: Side-to-side difference (reproducibility) — The experienced examiner performed tests on 20 healthy subjects
  Groups: Examiner effect group
Diagnostic Test: Side-to-side difference (availability) — Two examiners performed the test on one healthy subject with both devices for ten consecutive days.
  Groups: Method effect group
Diagnostic Test: Side-to-side difference (Accuracy) — 200 ACL rupture and 200 healthy subjects were recruited as contrast to compare the accuracy of the devices in diagnosing ACL rupture.
  Groups: Equipment effectiveness group

SUMMARY:
We introduced an automatic knee arthrometer (AKA) and aimed to evaluate the repeatability and effectiveness thereof in diagnosing ACL rupture compared with the KT-2000.

DETAILED DESCRIPTION:
The AKA was compared to the KT-2000 at 134 N in this study, the anterior displacement and difference of both knees of every subject were measured. The first protocol was designed to evaluate examiner effect (level of experience) and contralateral-side effect (left or right knee) in a single healthy subject, ten times, on ten consecutive days. The second was to compare the stability in 20 healthy subjects, with a single experienced examiner. Third, we recruited 200 ACL rupture and 200 healthy subjects as contrast to compare the accuracy of the devices in diagnosing ACL rupture.

ELIGIBILITY:
Inclusion Criteria:

* patients with ACL rupture from our institution were included. All patients were diagnosed by sports medicine specialists based on clinical manifestation, combined with imaging examinations, and hospitalized for further surgery.

Exclusion Criteria:

* Patients aged <18 or >45 years, with combined multiple knee ligament injury combinations, and/or limited range of motion of the knee (unable to flex to 20-30°)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: one healthy subject was tested with both devices for ten consecutive days to estimate examiner effect； 20 healthy subjects were tested with both devices to determine the method effect； 200 medicine students volunteered as healthy subjects; each with pain-free knees in the last three months, and without a history of knee injury； 200 patients with ACL rupture from our institution were also included.
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Side-to-side difference （SSD） | within 3 months after ACL rupture
  Side-to-side difference （SSD）at 134 N

CONTACTS AND LOCATIONS:
Overall Officials: yingfang ao, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided